CLINICAL TRIAL: NCT05906433
Title: Optimal Anesthetic for Corticosteroid Injections for Knee Osteoarthritis.
Acronym: Injections
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Florida Orthopaedic Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI_ PAL_V3_ 8
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee injection; Knee osteoarthritis; corticosteroid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone Acetonide; Bupivacaine; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: At screening/baseline, informed consent will be obtained, demographics and medical history will be collected, patient x-ray will be reviewed/KL grade confirmed, narcotic use in last 6 months will be screened using E-FORCSE (Florida Prescription Drug Monitoring Program) database, inclusion and exclusion criteria will be assessed, and patient will be randomized into one of the study groups. We will only include patients who are receiving unilateral knee injections. Further, patient's baseline information on VAS Pain and current medication (analgesic or NSAID) will be collected. VAS Pain will be also collected immediately after the intervention and 2 minutes after the intervention, in addition to global perceived improvement score and AEs.
  The intervention in this study is intra-articular knee injection of synthetic corticosteroid (kenalog) and variable amount of anesthetic (0ml, 2ml or 4 ml of 0.25% bupivacaine).
Who Masked: Participant
Masking Description: The PI standard of care is to offer patients who complain of knee pain a corticosteroids injection regardless of patient participation in a study. A consent will be obtained prior the injection by a trained/qualified team member. Subjects will be randomly allocated to groups by concealed allocation. Randomization sequence between three groups will be created using Excel and will be further stratified by sex within each block, to ensure even distribution. A set of numbered envelopes will be created, with each having one unique group assigned. A staff member will assign an envelope with group assignment upon consent and record envelope number ID. The ARNP will open an envelope, administer injection based on the group assigned. The ARNP will prepare the medication to maintain the double blinded aspect of the study. The ARNP is trained and experienced with injections and has giving injections for several years. She will not be involved in the evaluations of the patient pre/post injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Kenalog with 0ml bupivacaine (Experimental): The intervention in this study is one intra-articular knee injection of synthetic corticosteroid (kenalog) and variable amount of anesthetic,0ml of bupivacaine. The patients will be randomized into this group.
  Interventions: Drug: Kenalog with bupivacaine Injection
- Kenalog with 4ml bupivacaine (Experimental): The intervention in this study is one intra-articular knee injection of synthetic corticosteroid (kenalog) and variable amount of anesthetic,4ml of bupivacaine. The patients will be randomized into this group.
  Interventions: Drug: Kenalog with bupivacaine Injection
- Kenalog with 0.25% bupivacaine (Experimental): The intervention in this study is one intra-articular knee injection of synthetic corticosteroid (kenalog) and variable amount of anesthetic,0.25% of bupivacaine. The patients will be randomized into this group.
  Interventions: Drug: Kenalog with bupivacaine Injection

INTERVENTIONS:
Drug: Kenalog with bupivacaine Injection — Indications, relevant for this study include Kenalog injection for knee pain from osteoarthritis or inflammatory arthritis. A single injection to a patient who has no known allergies to anesthetic or corticosteroids would be administered during a scheduled clinical visit.
  Other Names: Knee Injection; Corticosteroid Injection; Kenalog; Bupivacaine

SUMMARY:
To evaluate pain relief from corticosteroid injection with and without anesthetic as well as with variable volume of anesthetic. Pain relief will be measured using the VAS pain score at the time of the injection as well as several time points following the injection to capture pain relief longevity. The investigators intend to evaluate how well the patients tolerate corticosteroid mixtures without anesthetic as well as with different volumes of anesthetic. Primary measure will be the time from procedure when postoperative status is considered success (as measured by global perceived improvement score).

DETAILED DESCRIPTION:
Primary objective is to evaluate pain relief from corticosteroids, Kenalog without anesthetic as well as with different volumes of anesthetic. The investigators will measure the VAS pain score at the time of the injection as well as several time points following the injection. Additionally, the investigators will evaluate how long the injection provided pain relief for the patient.

The secondary intend is to evaluate how well the patients tolerate Kenalog mixtures without anesthetic as well as with different volumes of anesthetic by using the VAS pain scale.

The investigators hypothesize that patient with lower volume of injection will experience less pain during the procedure and that there will be no statistically significant difference in pain level between the study groups during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age and be able to consent for themselves.
2. OA grade Kellgren Lawrence Stage II or III.
3. Diagnosis of primary osteoarthritis.

Exclusion Criteria:

1. Patients with other forms of arthritis such as inflammatory arthritis.
2. History of narcotic use for the past 6 months.
3. Kellgren Lawrence arthritis grade 1 or 4.
4. Pregnant women and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Injection for Knee Pain | Prior to procedure (in office)
  Visual Analogue Scale (VAS)
Injection for Knee Pain | Immediate post procedure (in office)
  Visual Analogue Scale (VAS)
Injection for Knee Pain | 2 minutes post procedure (in office)
  Visual Analogue Scale (VAS)
Injection for Knee Pain | Day 1 post procedure (phone interview)
  Visual Analogue Scale (VAS)
Injection for Knee Pain | Day 14 post procedure (through EDC)
  Visual Analogue Scale (VAS)
Injection for Knee Pain | Day 42 post procedure (in office)
  Visual Analogue Scale (VAS)
Injection for Knee Pain | Day 84 post procedure (through EDC)
  Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Assessment of Knee Pain | Immediate Post-op (in office)
  Global Perceived Improvement
Assessment of Knee Pain | Day 1 post procedure (phone interview)
  Global Perceived Improvement
Assessment of Knee Pain | Day 42 post procedure (in office)
  Global Perceived Improvement
Assessment of Knee Pain | Day 84 post procedure (through EDC)
  Global Perceived Improvement

OTHER OUTCOMES:
Medications | Prior to procedure (in office)
  Review of Medications
Medications | Day 1 post procedure (phone interview)
  Review of Medications
Medications | Day 14 post procedure (through EDC)
  Review of Medications
Medications | Day 42 post procedure (in office)
  Review of Medications
Medications | Day 84 post procedure (through EDC)
  Review of Medications
Review of Adverse Events | Immediate post procedure (in office)
  Any issues with procedure
Review of Adverse Events | Day 1 post procedure (phone interview)
  Any issues with procedure
Review of Adverse Events | Day 42 post procedure (in office)
  Any issues with procedure
Review of Adverse Events | Day 84 post procedure (through EDC)
  Any issues with procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedard NA, Dowdle SB, Anthony CA, DeMik DE, McHugh MA, Bozic KJ, Callaghan JJ. Response to Letter to the Editor on "The AAHKS Clinical Research Award: What Are the Costs of Knee Osteoarthritis in the Year Prior to Total Knee Arthroplasty?". J Arthroplasty. 2018 Jan;33(1):307. doi: 10.1016/j.arth.2017.10.002. Epub 2017 Oct 10. No abstract available. PMID 29079170
- [Background] Blankstein M, Lentine B, Nelms NJ. Common Practices in Intra-Articular Corticosteroid Injection for the Treatment of Knee Osteoarthritis: A Survey of the American Association of Hip and Knee Surgeons Membership. J Arthroplasty. 2021 Mar;36(3):845-850. doi: 10.1016/j.arth.2020.09.022. Epub 2020 Oct 8. PMID 33616067
- [Background] Grishko V, Xu M, Wilson G, Pearsall AW 4th. Apoptosis and mitochondrial dysfunction in human chondrocytes following exposure to lidocaine, bupivacaine, and ropivacaine. J Bone Joint Surg Am. 2010 Mar;92(3):609-18. doi: 10.2106/JBJS.H.01847. PMID 20194319
- [Background] Smith MD, Wetherall M, Darby T, Esterman A, Slavotinek J, Roberts-Thomson P, Coleman M, Ahern MJ. A randomized placebo-controlled trial of arthroscopic lavage versus lavage plus intra-articular corticosteroids in the management of symptomatic osteoarthritis of the knee. Rheumatology (Oxford). 2003 Dec;42(12):1477-85. doi: 10.1093/rheumatology/keg398. Epub 2003 Jul 16. PMID 12867587
- [Background] Parker RD, Streem K, Schmitz L, Martineau PA; Marguerite Group. Efficacy of continuous intra-articular bupivacaine infusion for postoperative analgesia after anterior cruciate ligament reconstruction: a double-blinded, placebo-controlled, prospective, and randomized study. Am J Sports Med. 2007 Apr;35(4):531-6. doi: 10.1177/0363546506296313. Epub 2007 Jan 23. PMID 17244900